CLINICAL TRIAL: NCT01716247
Title: Comparison of Contrast Enhanced Mammography to Breast MRI in Screening Patients at Increased Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-214
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Women at Increased Risk for Developing Breast Carcinoma
Keywords: Mammography (CESM); MRI; Breast screening; 12-214

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- pts at risk for breast cancer (Experimental): Women at increased risk for breast cancer who are being referred for screening MRI will be offered and consented for CESM at the same time. The 2 examinations will be performed on the same day when at all possible and if not we will make every attempt to perform CESM before MRI. Patients with outside MRI performed within 30 days and of adequate quality will also be eligible for CESM.
  Interventions: Other: Mammography (CESM) and MRI

INTERVENTIONS:
Other: Mammography (CESM) and MRI — The study consists of the addition of a single contrast enhanced digital mammography examination (CESM) to the routine screening of a woman at increased risk for breast cancer who is also having a breast MRI. Breast MRIs will be read by the radiologist reading breast MRIs on any given day. CESM is a dedicated system, derived from a standard digital mammography unit modified to deliver the dual or multiple energy exposures and visualization of combined images after IV contrast administration. If the patient is having her routine mammogram within 30 days of her MRI, CESM can replace that mammogram Patients will be randomly assigned to one of the radiologists trained to interpret CESM. That radiologist will read the CESM blinded to the results of the breast MRI.This process will be monitored by the research assistant No radiologist will read both the breast MRI and CESM on the same patient.

SUMMARY:
The purpose of this study is to determine if Contrast Enhanced Spectral Mammography (CESM) will be able to detect smaller/earlier breast cancers as well as breast MRI can.

ELIGIBILITY:
Inclusion Criteria:

* Women considered at increased risk for developing breast carcinoma (those with a lifetime risk of >15%due to family history, genetic predisposition, prior radiation therapy to the chest, prior biopsy showing a high risk lesion, or personal history of breast cancer) that are being screened with breast MRI.
* Women who have a screening digital mammogram on the day of CESM or within 365 days prior

Exclusion Criteria:

* Women under 21.
* Pregnant or possibly pregnant.
* Women who have a contraindication to the intravenous use of iodinated - contrast agent (i.e., allergy to iodinated contrastor severely impaired renal function with a creatinine level > or = to 1.3).
* Women with breast implants.
* Women with pacemakers.
* Women with aneurysm clips that don't allow for MRI.
* Women too claustrophobic to undergo MRI.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
compare the sensitivity and specificity CESM | 1 year
  CESM to that of breast MRI in a population of women who are being screened because they are at increased risk for developing breast cancer. For this purpose a positive CESM test will be defined as a score of 4 or 5. We will use the existing MRI BIRADS system to score CESM images based on the characteristics of individual lesions and increased enhancement compared to the background. A positive MRI test will be defined by a BIRADs score of 4 or 5.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Jochelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/